CLINICAL TRIAL: NCT02776891
Title: A Feasibility Study of Gallium-68 Citrate PET to Detect Aberrant MYC Protein Expression in Diffuse Large B-Cell Lymphoma
Brief Title: A Feasibility Study of Gallium-68 Citrate PET to Detect Aberrant MYC Proto-Oncogene, BHLH Transcription Factor (MYC) Protein Expression in Diffuse Large B-Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unexpected dose production issues prevented study start up
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16251
Record Dates: First submitted 2016-05-17; First posted 2016-05-18 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma
Keywords: lymphoma; gallium citrate; PET
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma | interventions — gallium citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gallium citrate (Experimental): The patients will be organized into two cohorts. Cohort 1 will receive 10 mCi and will be imaged 4 and 6 hours post injection. Cohort 2 will receive 15 millicurie (mCi) and will be imaged 4 and 6 hours post injection. Cohort 2 will be imaged if the optimal protocol identified image quality from cohort 1 does not allow for the resolution of cancer lesions.
  Interventions: Drug: Gallium citrate

INTERVENTIONS:
Drug: Gallium citrate — Ga-68 citrate will be administered on an outpatient basis at the Center for Molecular and Functional Imaging at China Basin. It will be administered a single time point intravenously prior to PET imaging. The one-time nominal injected dose will be up to 15 mCi containing 10 - 25 μg Ga-68. A simultaneous MRI (PET/MRI) of the head will be used for attenuation correction and anatomic localization of gallium-68 citrate uptake and standardized uptake value (SUV) calculation.
  Other Names: Ga-68 citrate

SUMMARY:
This is a single center imaging study investigating the use of PET with 68Ga-citrate in patients with DLBCL or BCLU.

DETAILED DESCRIPTION:
This is a single center feasibility imaging study in patients with diffuse large B-cell lymphoma (DLBCL) or B-cell Lymphoma, Unclassifiable with features between DLBCL and Burkitt's (BCLU). Study participants will undergo PET/MRI of the whole body with 68Ga citrate.

The study will include at least 5 patients with double hit lymphoma and 5 patients with DLBCL with an additional 5 more patients as expansion once the dose level has been established. Patients with DLBCL will be included once an optimal dose level for the resolution of cancer lesions has been established.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed DLBCL or BCLU.

   * Double hit lymphoma, defined by positive cytogenetic/ fluorescence in situ hybridization (FISH) analysis for translocations involving myc and bcl2 or a double hit score of 2 by immunohistochemistry as described by Johnson et al.
   * DLBCL without myc translocation or overexpression by the above methods
2. Presence of palpable or radiographically measurable disease of at least 1.5 cm in longest dimension.
3. Available prior CT or PET/CT scan done in the last 8 weeks for comparison
4. Prior chemotherapy or radiation to the measurable lesion must be completed at least 14 days prior.
5. Adequate renal function with estimated creatinine clearance ≥50 mL/min (by the Cockcroft Gault equation)
6. No contraindications to MRI (e.g. pacemaker, aneurysm clips, severe claustrophobia)
7. Ability to sign a study-specific internal review board (IRB) approved consent prior to study entry. Patients must be able and willing to consent and undergo study procedures.
8. Age ≥18 years old

Exclusion Criteria:

1. Any serious and/or unstable pre-existing medical, psychiatric, or other medical condition that could interfere with subject's safety, provision of informed consent, or compliance with study procedures
2. Body weight over 300 pounds
3. Female patients who are pregnant or breast-feeding
4. Prior MRI with gadolinium performed <24 hours before the study scan
5. No red blood cell transfusion or iron administration by any route in the last 7 days
6. Prior hypersensitivity or intolerance to gadolinium or gallium citrate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Uptake of radiotracer in tumor tissue | 16 months
  To show evidence of specific uptake of the radiotracer in the tumor tissue compared to background. For exploratory radiotracer studies, this is typically defined as 1.5-2 fold increase in SUVmax in the tumor compared to mediastinal blood pool activity.

SECONDARY OUTCOMES:
Comparing Gallium citrate uptake | 16 months
  To compare 68Ga-citrate (standard uptake value, metabolic tumor volume) between patients with Double Hit Lymphoma (DHL) and with diffuse B-cell lymphoma without aberrant MYC expression

CONTACTS AND LOCATIONS:
Overall Officials: Michael Evans, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No